CLINICAL TRIAL: NCT03993717
Title: Safety and Immunogenicity of Recombinant Glycoprotein E Herpes Zoster Subunit (HZ/su) Vaccine in Renal Transplant Recipients
Brief Title: Solid Organ Transplant SHINGRIX
Status: Terminated | Type: Observational
Why Stopped: Due to personnel changes and COVID-19.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Associate Professor, Emory University
Other Study IDs: IRB00109207
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplant; Complications
Keywords: shingles vaccine; immune responses; Clinical Trials; Immunology; Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Three to six months post-transplant Group: Subjects in this arm will receive the SHINGRIX vaccine three to six months after kidney transplant
  Interventions: Biological: SHINGRIX
- Twelve to thirty-six months post-transplant Group: Subjects in this arm will receive the SHINGRIX vaccine twelve to thirty-six months after kidney transplant
  Interventions: Biological: SHINGRIX

INTERVENTIONS:
Biological: SHINGRIX — A single intramuscular injection of the FDA-approved recombinant glycoprotein E herpes zoster (HZ/su) vaccine will be administered in the deltoid muscle of the preferred arm
  Other Names: Zoster vaccine recombinant

SUMMARY:
This study will assess the immune responses to the recombinant, AS01-adjuvanted varicella zoster virus subunit (HZ/su) vaccine or SHINGRIX in immunosuppressed patients, particularly those who have received a renal transplant, and aim to better understand if the vaccine and perhaps other adjuvanted vaccines are safe in these patients.

30 participants will be divided into 2 groups, one group will receive the 1st out of 2 doses of the vaccine 3-6 months after transplant per standard of care and the second group will receive the 1st out of 2 doses of the vaccine 12-36 months after the transplant per standard of care.The duration of the study is 180 days.

DETAILED DESCRIPTION:
Shingles is a viral illness caused by the same virus that causes the chicken pox. Reactivation of this virus leads to shingles which is a painful blistering rash. Around 10% of organ transplant patients get shingles. This study will help us assess the safety and efficacy of a new shingles vaccine, SHINGRIX in Kidney Transplant patients. SHINGRIX is FDA approved for the prevention of shingles.

In this study, participants will be divided into 2 groups, one group will receive the 1st out of 2 doses of the vaccine 3-6 months after transplant per standard of care and the second group will receive the 1st out of 2 doses of the vaccine 12-36 months after the transplant per standard of care.

This research is conducted at the Emory University Hospital and Emory Clinics. Additionally follow up visits might also be conducted at the Emory Hope Clinic, the clinical arm of the Emory Vaccine Center.

Subjects will be identified through review of medical records or by referral from their healthcare providers. Subjects may also self-refer from the IRB approved recruitment flyers. Following identification/referral, a coordinator or recruiter will contact the subject and tell them about the study and see if he/she is interested. If the potential subject is interested, the recruiter will obtain an oral consent and prescreen them for the study using a screening checklist. Qualified subjects will be scheduled to come into the clinic and be fully consented and proceed with screening/enrollment.

Blood specimens will be collected and stored for the research study and for future use. Subjects can opt to have their information stored in a Hope Clinic database in order to contact them for other studies they may qualify for in the future. There are no other optional studies planned at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of informed consent and provision of written informed consent before any study procedures.
2. Capable of attending study visits according to the study schedule
3. Males or females greater than or equal to 50 years of age.
4. Oral temperature less than 38 C.
5. Are in general good health, as determined by medical history and targeted physical exam related to this history
6. Recent renal transplant (either 3-6 months or 12-36 months prior)
7. Have received maintenance immunosuppressive therapy for prevention of allograft rejection for a minimum of 30 days prior to the first vaccination
8. Have received an ABO compatible allogeneic renal transplant
9. Male subjects should agree not to contribute to conception of a child, including sperm donation, for the duration of the study.

Exclusion Criteria:

1. Have received any transplant in addition to renal transplant
2. Have an acute illness within 72 hours prior to vaccination
3. Have a severe medical condition as determined by the investigators
4. Have kidney disease related to any known immune/autoimmune phenomena including, but not limited to: systemic lupus erythematosus, glomerulonephritis (post-streptococcal, Goodpasture syndrome, granulomatosis with polyangitis, polyarteritis nodosa, etc.).
5. Be on systemic immunosuppressive agents aside from those related to their renal transplant
6. Have known HIV or primary immune deficiency
7. Have a known potential immune-mediated disorder (pIMD)
8. Have planned receipt of any unlicensed or investigational medications, biologics, or vaccines for the duration of subject study participation
9. Have a history of severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine
10. Have donated blood or blood products within 56 days before study vaccination and for the duration of the study
11. Have received the Shingrix or Zostavax injection previously
12. Have had Shingles in the past
13. Be of child-bearing potential
14. Have known recent exposure to wild-type varicella in the past 4 weeks
15. Have a history of severe reactions following other vaccinations

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid Organ Transplant kidney recipients
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Change in levels of Anti-gE antibody concentrations | Day 1, Day 61, Day 180
  Anti-gE antibody concentrations will be obtained via enzyme-linked immunosorbent assay (ELISA)
Change in number of subjects with a vaccine response for anti-gE antibody | Day 61, Day 180
  Vaccine response is defined as:
  * For initially seronegative subjects, antibody concentration at post-vaccination greater than or equal to (≥) 4 fold the cut-off for Anti-gE (4x97 milli-international units per milliliter [mIU/ml])
  * For initially seropositive subjects (defined as ≥ 97 mIU/ml), antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.

SECONDARY OUTCOMES:
Number of subjects with any related severe adverse events (SAEs) | Day 180
  Number of participants with SAEs from first vaccination until the end of the trial
Number of subjects with any grade 3 related adverse events (AEs) | Day 91
  Number of subjects with any grade 3 related AEs from each vaccination and until 15 days after each vaccination
Number of subjects with renal allograft rejection | Day 180
  Number of subjects with renal allograft rejection from first vaccination until the end of the trial
Number of subjects with changes in allograft function | Day 180
  Number of subjects with changes in allograft function from first vaccination until the end of the trial.
  Allograft function will be defined as increase in serum creatinine levels (≥ 1.25, ≥ 1.50, ≥ 1.75 or ≥ 2 fold increase)
Change in HLA antibody titers | Day 1, Day 15, Day 61, Day 75, Day 180
  HLA antibody titers will be measured and analyzed at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Hope Clinic, Atlanta, Georgia
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No